CLINICAL TRIAL: NCT03093064
Title: The Role of Inflammation in Brain and Cognitive Function in Mental Disorders
Brief Title: Inflammatory Response In Schizophrenia
Acronym: IRIS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: King's College London (Other)
Collaborators: South London and Maudsley NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 208083
Record Dates: First submitted 2017-02-23; First posted 2017-03-28 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Natalizumab

STUDY DESIGN:
Intervention Model Description: This is an experimental medicine study, the purpose of which is provide a mechanistic understanding of neuroinflammation in schizophrenia by investigating response to natalizumab (phase 1b).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Patient Group: Natalizumab (Experimental): Natalizumab 300mg, intravenous, once monthly, total of 3 doses
  Interventions: Drug: Natalizumab
- Patient Group: Placebo (Placebo Comparator): Saline, intravenous, once monthly, total of 3 doses
  Interventions: Other: Placebo: normal saline

INTERVENTIONS:
Drug: Natalizumab — Natalizumab is a humanized monoclonal antibody against the cell adhesion molecule α4-integrin, currently licensed for the treatment of multiple sclerosis and Crohn's disease.
  Other Names: Tysabri
  Arms: Patient Group: Natalizumab
Other: Placebo: normal saline — Normal saline, intravenous infusion
  Arms: Patient Group: Placebo

SUMMARY:
Schizophrenia affects a significant proportion of the population and current levels of understanding of the illness is inadequate to treat it effectively. Converging lines of evidence suggest that neuroinflammation occurs in schizophrenia, and specifically over-activity of brain-resident immune cells called microglia. It is however unclear whether activated microglia play a primary role in schizophrenia, or whether this is a secondary phenomenon of no pathophysiological significance. The investigators therefore plan to test the effect of a monoclonal antibody (natalizumab) on psychotic symptoms in a cohort of first episode psychosis patients.

DETAILED DESCRIPTION:
One of the key aims of the study is to determine if there is a relationship between change in imaging inflammation markers from baseline to follow-up and changes in other markers of inflammation over the same period. In September 2021, an open label arm for natalizumab was added to the study. The relationship between changes in imaging inflammation markers and changes in other markers of inflammation will be analysed within subjects including all patients who received natalizumab.

ELIGIBILITY:
Inclusion criteria:

1. Aged 18-50 years
2. Diagnosis of schizophrenia or other psychotic disorder (Diagnostic and Statistical Manual of Mental Disorders-5 (DSM-5);
3. Symptomatic, defined as one or more positive symptom >3 AND one or more negative symptom >3 on the Positive and Negative Syndrome Scale (PANSS);
4. No acute relapse and psychiatrically stable for >1 month before screening;

Exclusion criteria:

1. History of significant co-morbid CNS disorder (including significant head trauma or significant loss of consciousness, Parkinson's Disease, Epilepsy, Alzheimer's Dementia, Huntington's Disease).
2. Any absolute contraindications to natalizumab, as per natalizumab SPC
3. Current or recent (last 3 months) infection, or history of significant infection, or an immunocompromised state
4. Previous use of natalizumab or previous use of other monoclonal antibody.
5. Ongoing long-standing use of oral steroids or non-steroidal anti-inflammatory drugs.
6. Pregnancy and/or breast-feeding.
7. Substance dependence/abuse other than to cigarettes.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2023-06-15 (Actual); Study Completion 2023-08-07 (Actual)

PRIMARY OUTCOMES:
Change in Translocator Protein (TSPO) availability pre- and post-natalizumab or placebo administration | Baseline TSPO availability will be assessed at day -14 prior to first administration of natalizumab/placebo (day zero). TSPO availability will be re-assessed post administration of natalizumab/placebo at day +57(+14 days)
  TSPO availability assessed using Positron Emission Tomography (PET)

SECONDARY OUTCOMES:
Correlation of TSPO availability with brain functional measures at baseline. | Baseline combined PET/MRI scan will be performed at day -14 prior to administration of natalizumab/placebo (day zero)
  Both TSPO availability (as measured using PET imaging) and brain functional measures (as measured using functional magnetic resonance imaging and magnetic resonance spectroscopy) will be measured simultaneously using a combined PET/MRI scanner.
Correlation of cerebrospinal fluid (CSF) inflammatory markers with brain functional measures at baseline. | Baseline PET/MRI scan will be performed at day -14 prior to administration of natalizumab/placebo (day zero). CSF collection will be performed between the time points day -14 to day -1 prior to administration of natalizumab/placebo (day zero).
  Brain functional measures assessed using functional magnetic resonance imaging and magnetic resonance spectroscopy.
  CSF inflammatory markers: measurements of cytokine concentrations (e.g. C-reactive protein, Interleukin-6)
Correlation of blood inflammatory markers with brain functional measures at baseline. | Baseline PET/MRI scan will be performed at day -14 prior to administration of natalizumab/placebo (day zero). Blood collection will be performed between the time points day -14 to day -1 prior to administration of natalizumab/placebo (day zero).
  Brain functional measures assessed using functional magnetic resonance imaging and magnetic resonance spectroscopy.
  Blood inflammatory markers: measurements of cytokine concentrations (e.g. C-reactive protein, Interleukin-6)
Longitudinal change in TSPO availability correlated with longitudinal change in brain functional measures. | Baseline combined PET/MRI scan will be performed at day -14 prior to administration of natalizumab/placebo (day zero). Repeat combined PET/MRI scan will be performed at day +57(+14 days).
  Both TSPO availability (as measured using PET imaging) and brain functional measures (as measured using functional magnetic resonance imaging and magnetic resonance spectroscopy) will be measured simultaneously using a combined PET/MRI scanner. There will be two separate scans - before and after administration of natalizumab/placebo.

CONTACTS AND LOCATIONS:
Overall Officials: Oliver D Howes, Principal Investigator — King's College London
Locations (1):
- Institute of Psychiatry, Psychology and Neuroscience, King's College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mizuno Y, Carreira Figueiredo I, Pillinger T, Hindley G, Baxter L, Parmar S, Lobo MC, Donocik JG, Rosenzweig I, Gupta A, Callegari I, Jeljeli S, Dunn JT, Hammers A, Awais R, Sander K, Arstad E, Politis M, Schubert JJ, Veronese M, Turkheimer FE, Reis Marques T, Howes OD. Immune alterations in schizophrenia and the effects of a therapeutic antibody: a neuroimaging study. Brain. 2025 Dec 1:awaf455. doi: 10.1093/brain/awaf455. Online ahead of print. PMID 41326319